CLINICAL TRIAL: NCT01273233
Title: A Blinded, Randomized and Controlled Clinical Trial of An Inactivated Enterovirus Type 71 Vaccine in Healthy Adults
Brief Title: Safety of an Inactivated Enterovirus Type 71 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EV71-1001-Ia
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Infection; Viral, Enterovirus
MeSH Terms: conditions — Infections; Enterovirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: 200U EV71 vaccine (Experimental): 12 adults received 3 doses of 200U EV71 vaccine 14 days apart
  Interventions: Biological: Inactivated Enterovirus Type 71 Vaccine
- Group 2: 400U EV71 vaccine (Experimental): 12 adults received 3 doses of 400U EV71 vaccine 14 days apart
  Interventions: Biological: Inactivated Enterovirus Type 71 Vaccine
- Group 1: Placebo (Placebo Comparator): 6 adults received 3 doses of placebo 14 days apart
  Interventions: Other: Placebo
- Group 2: Placebo (Placebo Comparator): 6 adults received 3 doses of placebo 14 days apart
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Inactivated Enterovirus Type 71 Vaccine — A Sinovac EV71 vaccine contains inactivated EV71 virus, aluminum hydroxide, sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate and injection water. The EV71 vaccine is supplied in one mono-dose vial containing 0.5 mL of viral suspension with EV71 virus antigen of 200U and 400U (Elisa unit)
  Other Names: EV71 Vaccine
  Arms: Group 1: 200U EV71 vaccine; Group 2: 400U EV71 vaccine
Other: Placebo — Placebo is suspension with a little ivory precipitation, composition of which is aluminum hydroxide diluents.
  Other Names: EV71 Vaccine
  Arms: Group 1: Placebo; Group 2: Placebo

SUMMARY:
A blind, randomized and placebo-controlled clinical trial with Inactivated Enterovirus Type 71 Vaccines in healthy adults

DETAILED DESCRIPTION:
A total of 36 eligible subjects aged from 18 to 49 years will be enrolled in the study, they will be randomized to receive two different dosage of vaccine candidate or placebo to evaluate the safety of this vaccine in adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, aged from 18 to 49 years old. Health is determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator
2. Provided legal identification for the sake of recruitment.
3. Subjects are able to understand and sign informed consents.

Exclusion Criteria:

1. Histroy of Hand-foot-mouth Disease
2. Women of lactation, pregnancy or about to be pregnant in 60 days
3. Subject that has allergic history of vaccine, or allergic to any ingredient of vaccine
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Congenital malformations or developmental disorders, genetic defects, or severe malnutrition
6. Epilepsy, seizures or convulsions history, or family history of mental illness
7. Autoimmune disease or immunodeficiency, or parents, brothers and sisters have autoimmune diseases or immunodeficiency
8. History of asthma, angioedema, diabetes or malignancy
9. History of thyroidectomy or thyroid disease that required medication within the past 12 months
10. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
11. Asplenia, functional asplenia or any condition resulting in the absence or removal the spleen
12. Acute illness or acute exacerbation of chronic disease within the past 7 days
13. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
14. History of any blood products within 3 months
15. Administration of any live attenuated vaccine within 28 days
16. Administration of subunit or inactivated vaccines ,e.g., pneumococcal vaccine, or allergy treatment within 14 days
17. Axillary temperature > 37.0 centigrade before vaccination
18. Abnormal laboratory parameters before vaccination
19. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of the inactivated Enterovirus Type 71 Vaccine in adults by different doses | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan-ping Li, MD, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China

REFERENCES:
- [Derived] Li YP, Liang ZL, Gao Q, Huang LR, Mao QY, Wen SQ, Liu Y, Yin WD, Li RC, Wang JZ. Safety and immunogenicity of a novel human Enterovirus 71 (EV71) vaccine: a randomized, placebo-controlled, double-blind, Phase I clinical trial. Vaccine. 2012 May 9;30(22):3295-303. doi: 10.1016/j.vaccine.2012.03.010. Epub 2012 Mar 15. PMID 22426327